CLINICAL TRIAL: NCT01834573
Title: Impact of Physical Exercise on Quality of Life in Patients With Inflammatory Bowel Disease - a Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: runIBD
Record Dates: First submitted 2013-04-14; First posted 2013-04-18 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Quality of Life in Patients With Inflammatory Bowel Disease
Keywords: inflammatory bowel disease; IBD; quality of life; Inflammatory Bowel Disease Questionnaire
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Patients of the intervention arm receive a 10 week exercise program
  Interventions: Behavioral: physical exercise
- Control (No Intervention): Patients of the control arm do not participate in exercise

INTERVENTIONS:
Behavioral: physical exercise — 10 weeks physical exercise; three times a week
  Arms: Intervention

SUMMARY:
Patients with inflammatory bowel disease (IBD) suffer from a diminished quality of life compared to healthy adults. This is due to the chronic course of disease accompanied with diarrhea, stomach pains but also with psychological stress.

It is known that physical education may improve course of disease and quality of life in a multitude of diseases. These include coronary heart disease, malignancies and also depression. The investigators believe that sport is as effective supportive tool in improving quality of life in IBD patients. But data is lacking with regard to controlled randomized clinical trials. Because of the small amount of data available the investigators considered a feasibility study. Our hypothesis is that IBD patients will cope with moderate exercise. The investigators further suspect that these patients improve their quality of life compared with patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* proven colitis ulcerosa (CU)
* proven crohns disease (CD)
* diagnosis >= 1 year before start of the study
* low or moderate disease activity

Exclusion Criteria:

* < 18 years
* high disease activity
* regular exercise > 2 hours per week
* diagnosis of CU oder CD < 1 year before start of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Quality of life | 10 weeks

SECONDARY OUTCOMES:
disease activity | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Klare, MD, Principal Investigator — II. Medizinische Klinik, Klinikum rechts der Isar München, Germany; Wolfgang Huber, MD, Study Director — II Medizinische Klinik, Klinikum rechts der Isar München, Germany
Locations (1):
- Klinikum rechts der Isar, München, Bavaria, Germany